CLINICAL TRIAL: NCT01481584
Title: Comparison of the Bioavailability the of a Single Administration of Two Canola Proteins (Hydrolyzate, Isolate) and Soy Protein in Healthy Men.
Brief Title: Nutritional Evaluation of Canola Protein in Comparison With Soy Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr., University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: LSEP H43-10
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Men
Keywords: Dietary protein; Canola protein; Protein metabolism; Protein-enriched drinks; Nitrogen balance
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — cyclopropapyrroloindole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Canola protein (Experimental): Canola protein (Brassica juncea; incorporated in a drink)
  Interventions: Dietary Supplement: Protein drink - protein isolate; Dietary Supplement: Protein drink - protein hydrolyzate
- Reference protein (Active Comparator): Reference Protein (soy protein isolate; incorporated in a drink)
  Interventions: Dietary Supplement: Protein drink - protein isolate; Dietary Supplement: Protein drink - protein hydrolyzate
- Wash out (No Intervention): Wash out (four weeks without any intervention between interventional periods)
- Run-in (No Intervention): Run-in period (three days before intervention, defined diet)

INTERVENTIONS:
Dietary Supplement: Protein drink - protein isolate — The subjects consumed 500 mL of a protein drink (tomato juice) containing 30 g protein (canola protein isolate or reference protein) after overnight fasting. After run-in period, each volunteer have to pass both protein-intervention days in different order with a four-week wash out period in between.
  Other Names: CPI
  Arms: Canola protein; Reference protein
Dietary Supplement: Protein drink - protein hydrolyzate — The subjects consumed 500 mL of a protein drink (tomato juice) containing 30 g protein (canola protein hydrolyzate or reference protein) after overnight fasting. After run-in period, each volunteer have to pass both protein-intervention days in different order with a four-week wash out period in between.
  Other Names: CPH
  Arms: Canola protein; Reference protein

SUMMARY:
The objective of the study is to evaluate the nutritional and physiological properties of two canola proteins focusing on the bioavailability in humans.

DETAILED DESCRIPTION:
The physiological effects of a single administration of two different industrially manufactured canola proteins (hydrolyzate, isolate) were investigated compared to soy protein.

Twenty-eight healthy men (ø 25 years) completed a double-blind, placebo-controlled, crossover study. The subjects were randomly divided into two groups (group A: canola protein isolate and soy protein isolate and group B: canola protein hydrolyzate and soy protein isolate). After a three-day run-in period, on the intervention day, the subjects consumed a protein drink containing 30.0 g protein powder added to a final volume of 500 mL tomato juice. Half of the subjects in each group consumed a protein drink containing 30.0 g canola protein, the other half received the soy protein. After taking of fasting blood samples in the morning of the intervention day, blood samples were drawn at regular intervals for a period of eight hours. At the end of the run-in period and on the intervention day, a 24-hour urine collection took place.

Within a second experiment (after 4 weeks), the protein source was crossed within the four subgroups for the second intervention.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker
* Body mass index: 20-26 kg/m²

Exclusion Criteria:

* Intake of pharmaceuticals
* Allergy against canola protein or soy protein
* Kidney disease

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Plasma amino acids | At Day 1 (Intervention day); After 0, 30, 60, 90, 120, 180, 240, 300, 360, 420 and 480 minutes
  Free proteinogenic amino acids

SECONDARY OUTCOMES:
Body composition (body status) | At day 1
  Bioelectrical impedance analysis, body weight
Nitrogen balance | After day 0 and 1
  Nitrogen balance = nitrogen intake - nitrogen output (urine nitrogen + fecal nitrogen + skin nitrogen); Nitrogen intake was calculated from food uptake; Urine nitrogen contains urea, uric acid, creatinine and total protein; Fecal nitrogen was calculated as the tenth part of the nitrogen intake; Skin nitrogen was calculated as 5.00 mg per kg of body weight

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutritional Physiology
Locations (1):
- Friedrich Schiller University Jena, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Fleddermann M, Fechner A, Rossler A, Bahr M, Pastor A, Liebert F, Jahreis G. Nutritional evaluation of rapeseed protein compared to soy protein for quality, plasma amino acids, and nitrogen balance--a randomized cross-over intervention study in humans. Clin Nutr. 2013 Aug;32(4):519-26. doi: 10.1016/j.clnu.2012.11.005. Epub 2012 Nov 14. PMID 23260747